CLINICAL TRIAL: NCT02141308
Title: Evaluation of the Utility of OCT Angiography in Assessing Vascular Perfusion in Rare Retinal and Choroidal Diseases
Brief Title: OCT in Rare Chorioretinal Diseases
Status: Recruiting | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Huang, Thomas Hwang, MD, Professor of Ophthalmology, Retina & Vitreous Diseases Division, Oregon Health and Science University
Other Study IDs: IRB00010511
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Retinal Artery Occlusions; Polypoidal Choroidal Vasculopathy; Retinal Arterial Macroaneurysm; Juxtafoveal Telangiecasia; Central Serous Chorioretinopathy
Keywords: Retina; Optical coherence tomography; Imaging
MeSH Terms: conditions — Retinal Artery Occlusion; Polypoidal Choroidal Vasculopathy; Retinal Arterial Macroaneurysm; Central Serous Chorioretinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Rare Chorioretinal Disease: Up to 150 patients diagnosed with a rare retinal or choroidal disease will be considered and evaluated for enrollment in this study.

SUMMARY:
This study will evaluate the total blood flow in the retina and choroid (structures in the back of the eye) by Doppler optical coherence tomography (OCT) and OCT angiography. Angiography is mapping of the blood vessels.

The purpose of measuring blood flow in the retina and choroid is to 1.) determine if rare diseases in these structures causes a change in blood flow compared to healthy eyes and 2.) find out if areas of changed blood flow line up with areas of damage that appear on conventional testing.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) is an imaging technology that can perform non-contact cross-sectional imaging of retinal and choroidal tissue structure in real time by measuring the intensity of reflected light. Tomographic images are generated by scanning the optical probe beam across the tissue structure of interest. OCT has become one of the most widely used imaging technologies by ophthalmologists. Its advantages include being a non-contact imaging modality, having micron-level resolution, producing a digital image that can be viewed electronically, and providing a reproducible quantitative measurement. New functional OCT including Doppler OCT and OCT angiography may allow an assessment of retinal blood flow and do away with the need for the more invasive fluorescein angiography (FA) test.

Thus, if the diagnostic data provided by functional OCT are at least equivalent or superior to those achieved by FA, patients and healthcare providers could realize a substantial benefit in utilizing this technology in the evaluation of retinal vascular disease. Even in the scenario in which an FA is not usually clinically indicated, OCT angiography may provide information over that of standard OCT and clinical examination and history, that might help clinicians better understand the etiology of the disease, and may even help inform treatment response.

ELIGIBILITY:
Subject-Level Criteria:

Inclusion a. Diagnosis of retinal or choroidal disease

Exclusion

1. Inability to give informed consent.
2. Inability to complete study tests within a 30 day period
3. Significant renal disease, defined as a history of chornic renal failure requiring dialysis or kidney transplant.
4. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g. unstable medical status including blood pressure, cardiovascular disease, and glycemic control).
5. Blood pressure > 180/110 (systolic above 180 OR diastolic above 110). If blood pressure is brought below 180/110 by anti-hypertensive treatment, subject can become eligible.
6. Women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months due to unknown safety of fluorescein angiography.

Study-Eye Criteria:

Inclusion

a. Diagnosis of retinal or choroidal disease

Exclusion

1. Inability to maintain stable fixation for OCT imaging.
2. An ocular condition is present that, in the opinion of the investigator, might affect or alter visual acuity during the course of the study (i.e. cataract)
3. Substantial cataract that, in the opinion of the investigator, is likely to decrease visual acuity by 3 lines or more (i.e. cataract would be reducing acuity to 20/40 or worse if the eye was otherwise normal).
4. Media opacity or otherwise that would prevent either fixation or ability to obtain adequate images as determined by the examiner.

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals 18 years of age and older presenting to the Retina Service within the Department of Ophthalmology at the Casey Eye Institute of Oregon Health & Science University with signs and symptoms of rare choroidal or retinal diseases will be evaluated for enrollment into this study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total Retinal and Choroidal Blood Flow | One year
  Determination whether disease affecting the retina and/or choroid shows a change in blood flow that differs from healthy eyes. Total retinal/choroidal blood flow will be measured in uL/min.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hwang, MD, Principal Investigator — Oregon Health & Science Univeristy
Locations (1):
- Casey Eye Institute, Oregon Health & Science University, Portland, Oregon, United States